CLINICAL TRIAL: NCT02829541
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single-Ascending-Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of BIIB068, a Bruton's Tyrosine Kinase Inhibitor, in Healthy Subjects
Brief Title: A Phase 1, Single-Ascending-Dose, Safety, Tolerability, Pharmacokinetic(PK), and Pharmacodynamic(PD) Study of BIIB068 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 236HV101
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Systemic Lupos Erythematosus, SLE
Keywords: Single Ascending Dose (SAD), Healthy Volunteers
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Agammaglobulinaemia Tyrosine Kinase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohorts 1 (Experimental): 6 participants randomized (4:2) to receive a single-ascending dose (SAD) administered orally in tablet
  Interventions: Drug: BIIB068; Drug: Placebo
- Cohort 2 (Experimental): 6 participants randomized (4:2) to receive a SAD administered orally in tablet(s)
  Interventions: Drug: BIIB068; Drug: Placebo
- Cohort 3 (Experimental): 8 participants randomized (6:2) to receive a SAD administered orally in tablet(s)
  Interventions: Drug: BIIB068; Drug: Placebo
- Cohort 4 (Experimental): 8 participants randomized (6:2) to receive a SAD administered orally in tablet
  Interventions: Drug: BIIB068; Drug: Placebo
- Cohort 5 (Experimental): 8 participants randomized (6:2) to receive a SAD administered orally in tablet(s)
  Interventions: Drug: BIIB068; Drug: Placebo
- Cohort 6 (Experimental): 14 participants (all active) to receive a SAD administered orally in tablet(s)
  Interventions: Drug: BIIB068

INTERVENTIONS:
Drug: BIIB068 — Administered as specified in the treatment arm.
  Other Names: Bruton's tyrosine kinase (BTK)
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohorts 1

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single oral doses of BIIB068 in healthy participants. Secondary objectives are to characterize the single-oral-dose Pharmacokinetic (PK) of BIIB068 in healthy participants, to determine the effect of food on the single-oral-dose PK of BIIB068 in healthy participants and to examine the effect of administration of the proton pump inhibitor (PPI) esomeprazole on the single-dose PK of BIIB068 in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* All male subjects must practice highly effective methods of contraception during the study and be willing and able to continue contraception and not donate sperm for at least 1 spermatogenic cycle (90 days) after administration of last dose of study treatment.
* All female subjects of childbearing potential must practice highly effective methods of contraception during the study and be willing and able to continue contraception for at least 1ovulatory cycle (30 days) after their last dose of study treatment.
* Must have a body mass index (BMI) between 18 and 32 kg/m2
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal (GI), hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of severe allergic or anaphylactic reactions, or history of any allergic reactions that in the opinion of the Investigator is likely to be exacerbated by any component of the study treatment.
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening or Day-1.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 9 Days Post dose
Number of participants with clinically significant laboratory assessment abnormalities | Up to 9 Days Post dose
Number of participants with clinically significant Vital sign abnormalities | Up to 9 Days Post dose
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | Up to 9 Days Post dose
Number of participants with clinically significant physical examination abnormalities | Up to 9 Days Post dose

SECONDARY OUTCOMES:
PK Assessment - Area Under the concentration-time curve from time zero to time of the Last Measurable Concentration (AUC0-tlast) | Up to 48 Hours Post dose
PK Assessment - Area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to 48 Hours Post dose
PK Assessment - Maximum observed concentration (Cmax) | Up to 48 Hours Post dose
PK Assessment - Time to reach maximum observed concentration (Tmax) | Up to 48 Hours Post dose
PK Assessment - Terminal elimination half-life (t1/2) | Up to 48 Hours Post dose
PK Assessment - Apparent total body clearance (CL/F) | Up to 48 Hours Post dose
PK Assessment - Apparent volume of distribution (Vz/F) | Up to 48 Hours Post dose
PK Assessment - Amount of BIIB068 excreted in urine (Aeu) | Up to 48 Hours Post dose
PK Assessment - Percentage (%fe) of BIIB068 excreted in urine | Up to 48 Hours Post dose
PK Assessment - Renal clearance (CLr) | Up to 48 Hours Post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Evansville, Indiana, United States